CLINICAL TRIAL: NCT02504450
Title: Outcomes of Antipsychotic Medication Use in the Emergency Department: A Retrospective Comparison Study
Brief Title: Outcomes of Antipsychotic Medication Used in the Emergency Department
Acronym: OAMED
Status: Completed | Type: Observational
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Other Study IDs: AHC6066
Record Dates: First submitted 2015-07-17; First posted 2015-07-22 (Estimated); Last update posted 2024-10-04 (Actual); Status verified 2016-07

CONDITIONS: Agitation,Psychomotor
Keywords: Bipolar 1 disorder; schizophrenia
MeSH Terms: conditions — Psychomotor Agitation; Schizophrenia | interventions — Loxapine; Haloperidol; ziprasidone

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Adasuve — Inhaled medication to treat acute agitation in the emergency department
  Other Names: Loxapine
Drug: Alternative medications — Medication given to treat acute agitation in the emergency department
  Other Names: Haloperidol, Serenace, Peridol, Haldon, Geodon, Ziprasidone

SUMMARY:
To review records of patients treated with antipsychotics (including Adasuve, Geodon, Haldol) in order to evaluate outcomes.

DETAILED DESCRIPTION:
A retrospective chart review will be performed for all patients presenting to the ED with agitation and subsequently given antipsychotic therapy for treatment. Identification of patients will be through chart review of patients presenting with agitation. Data to be recorded include patient age, gender, medical history, time of presentation, time of treatment, co morbidities, use of restraint, time to disposition and patient outcome. Inclusion criteria include all patients over age 18 presenting to the ED with agitation and treated with antipsychotics. No patients will be knowingly excluded from analysis. We will compare resulting outcomes of patients treated for agitation to see if Adasuve is superior to other commonly prescribed antipsychotics through its rate of discharge home and overall time in the emergency department.

ELIGIBILITY:
Inclusion Criteria:

* All patients given antipsychotic therapy for acute agitation

Exclusion Criteria:

* None

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: subjects treated in the emergency department for agitation
Sampling Method: Probability Sample
Enrollment: 93 (Actual)
Dates: Start 2015-04; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Length of stay in the emergency department | Participants will be followed for the duration of emergency department stay, an expected average of 12 hours.
  We will compare resulting outcomes of patients treated for agitation to see if Adasuve is superior to other commonly prescribed antipsychotics through its rate of discharge home and overall time in the emergency department.

SECONDARY OUTCOMES:
Disposition | Participants will be followed for the duration of emergency department stay, an expected average of 12 hours.
  disposition (home, transfer, admit), and time to disposition

CONTACTS AND LOCATIONS:
Overall Officials: Erik Kulstad, MD, Principal Investigator — Advocate Healthcare

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Dinh KV, Myers DJ, Noymer PD, Cassella JV. In vitro aerosol deposition in the oropharyngeal region for Staccato loxapine. J Aerosol Med Pulm Drug Deliv. 2010 Aug;23(4):253-60. doi: 10.1089/jamp.2009.0814. PMID 20528148
- [Result] Valdes J, Shipley T, Rey JA. Loxapine inhalation powder (adasuve): a new and innovative formulation of an antipsychotic treatment for agitation. P T. 2014 Sep;39(9):621-3, 648. PMID 25210413